CLINICAL TRIAL: NCT06123247
Title: Mothers' Perception Of Respect/Mistreatment During Pregnancy & Childbirth In Assiut Governorate
Brief Title: Mothers' Respect/Mistreatment During Pregnancy & Childbirth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdelrahman Mohamed, doctor, Assiut University
Other Study IDs: 04-2023-200266
Record Dates: First submitted 2023-08-03; First posted 2023-11-08 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Childbirth Problems; Pregnancy Related
Keywords: respect; mistreatment; mothers

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pregnancy and childbirth are important events in a woman's and family's life and a time of great vulnerability for every country and culture on earth. Although the concept of "safe motherhood" is often limited to physical safety, the birth of a child is also an important life milestone for women and their familiesin our study for ssessing the degree of respectful maternity care, or mistreatment during pregnancy and childbirth in Assiut Governorate, Egypt and Exploring the factors associated with respectful maternity care and mistreatment among Egyptian women in Assiut governorate in rural and urban areas .

DETAILED DESCRIPTION:
A woman's experience with childbirth care is an important factor in her future decisions about whether to receive health care through a health care facility. Women's negative encounters with health workers long-term injury and emotional trauma can result during childbirth. Every woman has several rights. They include the following rights: 1- Freedom from harm and abuse, 2- Information, informed consent and refusal, and respect for women's choices and preferences, including companion during childbirth, 3- Privacy and confidentiality 4) Respectful and dignified treatment 5 - Equality, non-discrimination and appropriate care 6- Healthcare and attainable high standards of health and 7- Freedom, autonomy, self-determination and non-coercion. Reported forms of disrespect and abuse fell into seven categories: physical abuse, non-consensual care, non-confidential care, indecent care, discrimination based on patient characteristics, abandonment of care, and incarceration in institutions.. RMC focuses on eliminating unhealthy and abusive behaviors by healthcare providers and associated personnel, and providing a sensitive and encouraging work environment to help women feel satisfied during childbirth.To measure women's experience of respectful maternity care, vedam et la developed Mothers on Respect Index (MORi) assesses the nature of patient-provider interactions and their impact on human feelings of respect during obstetric care .The mistreatment index (MIST index), which is an indicator of abuse consistent with the seven dimensions ( physical abuse, sexual abuse, verbal abuse, stigma and discrimination. Failure to meet professional standards of care, poor rapport during interactions with Providors, and the poor state and limitations of the healthcare system )

ELIGIBILITY:
Inclusion Criteria:

Women who have delivered (either vaginally or cesarean) in the past 8 weeks.

Exclusion Criteria:

* Women who had complicated childbirth, or stillbirth/neonatal death during their Last delivery will be excluded. In addition, women with known psychiatric illness . These women will be excluded . women who refuse to participate in the study will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: study will be conducted in two urban and two rural maternity and child health centers selected randomly from Assiut governorate We will recruit women who have given birth (either vaginal or Cesarean deliveries) within 8 weeks since their Last delivery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
measurement the degree of respectful maternity care, or mistreatment during pregnancy and childbirth in Assiut Governorate, Egypt | within 8 weeks after childbirth
  questionnaire including mothers of respect index and mistreatment index

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud zakhira, professor, Study Director — obstetrics &gynacology depatmen ,assiut university; moustfa alsonbaty, doctorate, Study Chair — obstetrics & gynacology depatmen assiut university
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Housseine N, Rijken MJ, Punt MC, Meguid T, Franx A, van der Graaf R, Browne JL. Mistreatment during childbirth. Lancet. 2020 Sep 19;396(10254):816-817. doi: 10.1016/S0140-6736(20)31556-7. No abstract available. PMID 32950087
- [Background] Vogel JP, Bohren MA, Tuncalp Ӧ, Oladapo OT, Gulmezoglu AM. Promoting respect and preventing mistreatment during childbirth. BJOG. 2016 Apr;123(5):671-4. doi: 10.1111/1471-0528.13750. Epub 2015 Dec 1. No abstract available. PMID 26628382
- [Background] Galle A, Manaharlal H, Cumbane E, Picardo J, Griffin S, Osman N, Roelens K, Degomme O. Disrespect and abuse during facility-based childbirth in southern Mozambique: a cross-sectional study. BMC Pregnancy Childbirth. 2019 Oct 22;19(1):369. doi: 10.1186/s12884-019-2532-z. PMID 31640603
- [Background] Savage V, Castro A. Measuring mistreatment of women during childbirth: a review of terminology and methodological approaches. Reprod Health. 2017 Oct 26;14(1):138. doi: 10.1186/s12978-017-0403-5. PMID 29073914